CLINICAL TRIAL: NCT04115995
Title: Perforator Mapping and Anastomosis Patency Evaluated by Dynamic Fluorescence Video Angiography of Indocyanine Green and Infrared Thermography.
Brief Title: DIEP Flap Perfusion Evaluated by DIRT and ICG-FA.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 22017/1641
Record Dates: First submitted 2019-04-16; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2018-12

CONDITIONS: Reconstructive Surgical Procedures
Keywords: Breast reconstruction; Perforator flaps; Computer Tomography; Indocyanine green; Fluorescence angiography; Infrared thermography; Dynamic infrared thermography; Doppler ultrasound; Angiosome; Perforasome; Flap perfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dynamic infrared thermography (DIRT) and indocyanine green fluorescence angiography (ICG-FA) — DIRT and ICG FA are used intraoperatively to evaluate perfusion of the perforators and the anastomosis. Both technique are compared in their ability to visualize perfusion.

SUMMARY:
Patients selected for DIEP breast reconstruction were examined with preoperative CTA, Doppler Ultrasound, dynamic infrared thermography (DIRT) and Indocyanin green fluorescent angiography (ICG-FA) for perforator mapping. DIRT and ICG-FA were used to evaluate perfusion of selected perforators. Following anastomoses for the DIEP flap to internal mammary vessels , patency of the anastomosis was evaluated with DIRT and ICG-FA. Recorded images from all the modules were compared.

DETAILED DESCRIPTION:
Introduction:

'The primary aim of our study is to compare invasive and non-invasive techniques to select a dominant perforator when harvesting a DIEP-flap for autologous breast reconstruction.

The secondary aim is to compare Dynamic Infrared Thermography (DIRT) and Laser Fluorescence Angiography (LFA) of Indocyanine green (ICG) in order to see whether they could be useful in the early detection of insufficient perfusion following the microvascular anastomotic procedure in DIEP flaps.

Material and Method:

Patients selected for breast reconstruction with autologous tissue were examined with preoperative CTA and a handheld Doppler Ultrasound for perforator mapping. Thereafter visual images from same area was obtained with dynamic infraredeed thermography (DIRT) and Indocyanin green fluorescent angiography (ICG-FA) before and after dissection of the skin flap with preserved medial and lateral DIEP perforators. Reconstructed breasts with hemi-DIEP-flaps were intraoperatively evaluated with DIRT and LFA immediately after the completion and opening of the microvascular anastomosis.The recorded images from the different techniques were assesses in relation to clinical outcome.

.

ELIGIBILITY:
Inclusion Criteria:

* Post mastectomy.
* Previously breast cancer patent treated with radiation therapy.
* Breast implant reconstruction is not possible or undesired.
* Healthy patient with moderate amounts of abdominal skin laxity.
* Patient who requires a minimal to moderate volume breast reconstruction.
* The patient willing to undergo the long, complex procedure and prolonged postoperative recovery.
* The patient willing to accept an abdominal scar and a potential for donor site morbidities.
* Patients operated with prophylactic salpingo-oophorectomy due to BRCA gene mutation.

Exclusion Criteria:

* Pregnancy and lactation.
* Patents below the age of 18 year.
* Renal failure or hepatic failure.
* Previous allergic reactions to ICG and iodide.
* Abdominal donor site that cannot be closed primarily.
* Previous TRAM flap or abdominoplasty.
* Significant medical comorbidities that make the patient a poor surgical candidate.
* Sigarette smoking or snuff.
* Obesity / BMI > 30.
* Previous abdominal suction-assisted lipectomy.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients are included for breast reconstruction after treatment for breast cancer.
Study Population: Female patients selected for autologous breast reconstruction with a DIEP flap.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-12-24 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of quality and location of perforating blood vessels with dynamic infrared thermography and indocyanine green angiography in autologous breast reconstruction: A comparative imaging study. | 2 year
  Pre-and intraoperative use of two different imaging technologies to assess quality and location of perforating blood vessels in autologous breast reconstruction. In this study we will compare images obtained using a non-invasive imaging technique, dynamic infrared thermography and an invasive imaging technique, laser fluorescence angiography of indocyanine green.
Quality of microvascular anastomosis by measuring perfusion through the anastomosis using dynamic infrared thermography and laser fluorescence angiography of indocyanine green. | 2 years
  The microvascular anastomosis provides blood supply to tissue used in breast reconstruction. The blood flow through the microvascular anastomosis can be monitored by use of different imaging techniques. In this study, perfusion images obtained by non-invasive dynamic infrared thermography and invasive fluorescence angiography of indocyanine green will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity Hospital of North Norway, Tromsø, Norway